CLINICAL TRIAL: NCT02164175
Title: Data Collection Registry of the HeRO Graft for End Stage Renal Disease Patients Receiving Hemodialysis
Status: Withdrawn | Type: Observational
Why Stopped: Company acquired and trial was not pursued
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HRG1301.000-M
Record Dates: First submitted 2014-05-29; First posted 2014-06-16 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: HeRO Graft

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HeRO Graft: End stage renal disease patients who receive HeRO Graft implant for dialysis access
  Interventions: Device: HeRO Graft implant for dialysis access

INTERVENTIONS:
Device: HeRO Graft implant for dialysis access — End Stage Renal Disease patients who receive HeRO Graft implant for dialysis access

SUMMARY:
Data Collection Registry of the HeRO Graft for End Stage Renal Disease Patients Receiving Hemodialysis

DETAILED DESCRIPTION:
Data collection including medical history, operative procedure data, and follow-up data every six months while using the HeRO Graft for dialysis, including:

* Post-operative complications for HeRO Graft implantation
* Length of time between insertion and use of HeRO Graft
* Incidence of thrombosis
* Hospitalizations
* Incidence of infections and other adverse event occurrence
* Mortality
* Hemoglobin
* Kt/V
* pre-dialysis blood pressure
* post-dialysis blood pressure
* blood flow rate and
* dialysis flow rate

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for HeRO Graft for dialysis access
* Age greater than 18 years old
* Able to give informed consent

Exclusion Criteria:

* Subjects with any kind of disorder that compromises the ability of the subject to give informed consent and/or to comply with the study procedures;
* Any medical condition that in the opinion of the investigator may pose a safety risk to a subject in the study or which may interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible for HeRO Graft for dialysis access
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the death rate of participants using the HeRO Graft is less than the death rate of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.

SECONDARY OUTCOMES:
Adequacy of dialysis (Kt/V) | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the adequacy of dialysis of participants using the HeRO Graft is better than the adequacy of dialysis of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.
Infection rate | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the infection rate of participants using the HeRO Graft is less than the infection rate of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.

OTHER OUTCOMES:
Hospitalization rate | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the hospitalization rate of participants using the HeRO Graft is less than that of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.
Patency rate | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the patency rate of participants using the HeRO Graft is less than that of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.
Intervention rate | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the intervention rate of participants using the HeRO Graft is less than that of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.
Adverse events | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the number of adverse events of participants using the HeRO Graft is less than that of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.
Blood pressure | Every six months post-implant until death or no longer using HeRO Graft for dialysis, up to five years
  To evaluate if the blood pressure of participants using the HeRO Graft is less than that of patients who do not receive the HeRO Graft and continue to use a tunneled dialysis catheter for dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lawson, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - Baylor Research Institute, Dallas, Texas
  - Sentara Medical Group Sentara Vascular Specialists, Norfolk, Virginia

REFERENCES:
- [Background] Gage SM, Katzman HE, Ross JR, Hohmann SE, Sharpe CA, Butterly DW, Lawson JH. Multi-center experience of 164 consecutive Hemodialysis Reliable Outflow [HeRO] graft implants for hemodialysis treatment. Eur J Vasc Endovasc Surg. 2012 Jul;44(1):93-9. doi: 10.1016/j.ejvs.2012.04.011. Epub 2012 May 12. PMID 22580402
- [Background] Katzman HE, McLafferty RB, Ross JR, Glickman MH, Peden EK, Lawson JH. Initial experience and outcome of a new hemodialysis access device for catheter-dependent patients. J Vasc Surg. 2009 Sep;50(3):600-7, 607.e1. doi: 10.1016/j.jvs.2009.04.014. Epub 2009 Jul 22. PMID 19628360
- [Background] Nassar GM, Glickman MH, McLafferty RB, Croston JK, Zarge JI, Katzman HE, Peden EK, Lawson JH, Martinez JM, Thackeray L. A comparison between the HeRO graft and conventional arteriovenous grafts in hemodialysis patients. Semin Dial. 2014 May-Jun;27(3):310-8. doi: 10.1111/sdi.12173. Epub 2014 Jan 15. PMID 24428351
- See also: HeRO Graft website — http://www.herograft.com